CLINICAL TRIAL: NCT03327896
Title: The Impact of Patient Complexity on Healthcare Utilization
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: OCHIN, Inc. (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: HSD-1603-34987
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Primary Care Quality Metrics; Well Child Visits in First 15 Months of Life NQF 1392; Diabetes Mellitus NQF 0059; Colorectal Cancer Screening NQF 0034; Emergency Department Utilization; Alcohol and Drug Screening
Keywords: Quality Measures, Social Determinants of Health

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- OCHIN EHR: Patients who were established patients at OCHIN Primary Care Clinics in 2015 and had a face to face visit at the clinic in 2015.
  Inclusion criteria for specific outcomes varies by criteria for demoninator specification for the metric.
  Interventions: Other: Charlson score and Community Social Deprivation
- OneFlorida EHR: Patients who were established patients at OneFlorida Primary Care clinics in 2015 and had a face to fact visit at the clinic in 2015.
  Inclusion criteria for specific outcomes varies by criteria for demoninator specification for the metric.
  Interventions: Other: Charlson score and Community Social Deprivation
- Oregon Medicaid: Clients who were continuously insured through Oregon Medicaid in 2015 and had a claim with an Evaluation and Management Current Procedure Terminology (CPT) code indicating an office visit listing a Primary Care provider as the performing provider.
  Inclusion criteria for specific outcomes varies by criteria for demoninator specification for the metric.
  Interventions: Other: Charlson score and Community Social Deprivation
- Florida Medicaid: Clients who were continuously insured through Florida Medicaid in 2015 and had a claim with an Evaluation and Management Current Procedure Terminology (CPT) code indicating an office visit listing a Primary Care provider as the performing provider. Florida Medicaid data is limited to clients who were 22 years or younger.
  Inclusion criteria for specific outcomes varies by criteria for demoninator specification for the metric.
  Interventions: Other: Charlson score and Community Social Deprivation

INTERVENTIONS:
Other: Charlson score and Community Social Deprivation — This is an observational study of the association of clinical comorbidity and neighborhood social deprivation characteristics with healthcare performance assessment.

SUMMARY:
Healthcare providers are routinely being assessed for metrics designed to assess the quality of the care they deliver. There is growing consensus that these measurements, which typically assess the percentage of patients meeting a specific standard of care, should be adjusted for the clinical complexity of the providers. This study will assess whether adjusting for the social complexity of the patient panel adds significantly to adjustment for clinical complexity in explaining apparent differences in quality of care provided by Primary care providers and clinics.

DETAILED DESCRIPTION:
The analysis will be conducted in 2 stages. In the first stage, indicators of social complexity (as assessed by characteristics of the patients' geocoded addresses) will be tested for significant association with patient level outcomes (meeting or not meeting a specific standard of care). These indicators will be assessed in 4 cohorts: 2 cohorts of patients identified in electronic health records of Clinical Research Networks of community health centers, and 2 cohorts of patients insured by Medicaid in 2015 (Oregon and Florida Medicaid cohorts). Due to limitations in the available data, some quality indicators can only be evaluated in a subset of the cohorts. The consistency of specific social complexity indicators, referred to as Community Vital Signs (CVS), will be evaluated across the cohorts and quality metrics.

In the second stage, CVS indicators that contributed consistently to models at the patient level will be evaluated for their effect on provider ranking on quality metrics if the metrics are adjusted for the social complexity of the providers' patient panel in addition to the panels' clinical complexity.

ELIGIBILITY:
Inclusion criteria for clinics: Clinics must be a clinic that offers Primary Care (Family Medicine Clinics, Pediatrics Clinics, General Practice Clinics, Internal Medicine clinics that are not limited to a subspecialty focus, and multi-specialty clinics that include primary care providers as part of a comprehensive care team.) Clinics must have implemented their EHR by 1/1/2014.

Inclusion criteria for patients: EHR Patients must be established patients within a health care system: at least one ambulatory visit to an included clinic in 2015 and at least 1 visit to a primary care clinic within the same health system prior to that visit.

Inclusion criteria for patients for Medicaid based Outcomes: Patient must have been continuously covered by Medicaid in 2015 and have had at least 1 visit billed as an office visit in 2015 with a provider identified as a primary care provider and at least 1 prior claim billed to the same provider. Patients must meet the age/condition criteria for the assessment of at least 1 secondary outcome.

Exclusion Criteria:

Exclusion criteria for patients: Patients with no geocoded address on file will be excluded from the analysis.

Exclusion criteria for patients for Medicaid based Outcomes: Patient with Medicaid coverage gaps of >45 days will be excluded from theses analyses. Exclusion criteria for providers: Providers with <20 patients in any Quality metric denominator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stage 1 (Patient Level): Established patients of primary care providers with a visit in 2015 Stage 2 (Provider level): Primary Care providers with at least 20 patients from established patients in 2015 Stage 3 (Clinic level): Primary care Clinics
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Provider Ranking as Assessed by Health Care Quality Metrics | 1 year (2015)
  Comparison of adjusted provider quality rankings with metrics adjusted for Charlson Morbidity Scores and Patient Panel Neighborhood Deprivation Indicators

SECONDARY OUTCOMES:
Well Child Visits in first 15 Months of life (patient level) | 15 months
  Number of well child visits in first 15 months of life in children turning 15 months in 2015
Screening for alcohol and drug misuse (patient level) | 1 year (2015)
  Documented screening for alcohol or drug misuse in patients aged 12 and over
Emergency Department Visits (Patient level) | 1 year (2015)
  Age stratified Emergency department visit rates in patients in Medicaid cohorts
Avoidable Emergency Department Visits (Patient level) | 1 year (2015)
  Age stratified Avoidable Emergency department visit rates in patients in Medicaid cohorts
Uncontrolled Hemoglobin A1c in Diabetics (patient level) | 1 year
  Last recorded HbA1c greater than 9 in patients with recorded diagnosis of Diabetes (EHR cohorts only)
Colorectal Cancer Screening (Patient level) | 1 year
  Documented colorectal cancer screening in 2015 (Oregon Medicaid cohort only)

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Sears, MBA, Principal Investigator — OCHIN, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hughes LS, Phillips RL Jr, DeVoe JE, Bazemore AW. Community Vital Signs: Taking the Pulse of the Community While Caring for Patients. J Am Board Fam Med. 2016 May-Jun;29(3):419-22. doi: 10.3122/jabfm.2016.03.150172. PMID 27170802
- See also: Article abstract — https://www.ncbi.nlm.nih.gov/pubmed/?term=27170802